CLINICAL TRIAL: NCT02841982
Title: Quadratus Lumborum Block : Effect on Acute Pain and Quality of Recovery After Laparoscopic Renal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cui Xulei (Other)
Responsible Party: Sponsor-Investigator, Cui Xulei, Attending physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: cuixulei3
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Laparoscopic Renal Surgery; Pain Management; Nerve Block
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- single-injection QLB(quadratus lumborum block) (Experimental): Single-injection of QLB is given preoperatively + postoperative IPCA(intravenous patient controlled analgesia)
  Interventions: Procedure: single-injection QLB(quadratus lumborum block); Device: Philip CX50 Ultrasound Scanner; Device: PAJUNK StimuLong; Drug: single dose ropivacaine; Drug: Morphine given as IPCA(intravenous patient controlled analgesia)
- IPCA (Active Comparator): postoperative IPCA is given alone
  Interventions: Drug: Morphine given as IPCA(intravenous patient controlled analgesia)

INTERVENTIONS:
Procedure: single-injection QLB(quadratus lumborum block) — Inject local anesthetics in between quadratus lumborum and psoas major without continuous local infusion
  Arms: single-injection QLB(quadratus lumborum block)
Device: Philip CX50 Ultrasound Scanner — The curved (C1-5) probe of Philip CX 50 Ultrasound Scanner is used for scan
  Arms: single-injection QLB(quadratus lumborum block)
Device: PAJUNK StimuLong
  Arms: single-injection QLB(quadratus lumborum block)
Drug: single dose ropivacaine — * 0.6ml/kg 0.5% ropivacaine with 1:200,000 adrenaline.
  * given immediately after the correct position of the tip of the needle has been verified.
  Arms: single-injection QLB(quadratus lumborum block)
Drug: Morphine given as IPCA(intravenous patient controlled analgesia) — bolus: 1.5~2mg, lock time: 10min, 1h limitation: 6~8mg

SUMMARY:
This prospective, randomized study,control study aims to compare the analgesic effect,opioids consumption,quality of recovery,length of hospital stay and incidence of chronic pain,et al. between single-injection QLB(quadratus lumborum block)+ intravenous patient-controlled analgesia (IPCA) and intravenous patient-controlled analgesia (IPCA) alone in patients undergoing laparoscopic renal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 yrs
* American Society of Anesthesiologists physical statusⅠ-Ⅲ
* Undergo laparoscopic nephrectomy
* Informed consent

Exclusion Criteria:

* A known allergy to the drugs being used
* Coagulopathy, on anticoagulants
* Analgesics intake, history of substance abuse
* Participating in the investigation of another experimental agent
* Inability to properly describe postoperative pain to investigators (eg, language barrier, neuropsychiatric disorder)

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
cumulative morphine consumption | within 48 postoperative hours

SECONDARY OUTCOMES:
The pain scores determined by the numeric rating scale (NRS, 0-10) | At 0, 2,4, 8, 12, 24 ,48,72hours after the surgery
nausea and vomiting score | within 24 hours after the surgery
pruritus score | within 24hour after the surgery
ambulation time | within the 7 days after surgery
time of recovery of bowl movement | within the 5 days after surgery
quality of recovery | 3days and 5days after surgery
  use the self-assessment 15 item QoR scale to assess the patient's recovery
Postoperative hospital length of stay | Up to 6 weeks
patient satisfaction with anesthesia | 48 hours after surgery
  use the Chinese version Bauer questionnaire to assess the patient satisfaction with anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, MD., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Xulei CUI, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No